CLINICAL TRIAL: NCT06947655
Title: Impact of Two Different Perioperative Tourniquets on Blood Loss, Surgical Field and Surgeon Satisfaction During Total Knee Arthroplasty
Brief Title: Impact of Different Perioperative Tourniquets on Blood Loss and Surgeon Satisfaction in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024_J
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The active control group receives a standarized FDA approved perioperative tourniquet (VBM-Tourniquet, VBM Medical, Sulz, Germany).
  Interventions: Device: VBM Tourniquet
- Intervention Group (Experimental): The intervention groups receives a standarized, FDA-approved perioperative tourniquet (Adaptive Cuff, Delfi Medical Innovations Inc., Vancouver, Canada).
  Interventions: Device: Adaptive Cuff

INTERVENTIONS:
Device: VBM Tourniquet — Perioperative VBM-Tourniquet Application with a fixation pressure of 15mmHg.
  Arms: Control
Device: Adaptive Cuff — Perioperative Delfi-Tourniquet Application with a fixation pressure of 15mmHg.
  Arms: Intervention Group

SUMMARY:
The present study investigates the impact of two different perioperative tourniquets with different closing features on operative blood los, surgical field quality and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Inidication for a Total Knee Arthroplasty
* Approval for Surgery by the Department of Anesthesia

Exclusion Criteria:

* Open Wounds of the lower extremities
* Acute or chronic infections of the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Loss | Perioperative
  Perioperative blood loss in ml.
Surgeon Satisfaction | Perioperative
  Surgical Satisfaction on a 0-100 mm VAS

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No